CLINICAL TRIAL: NCT02114801
Title: Mechanical Control of Plaque in Patients With Cerebral Palsy: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of the Valleys of Jequitinhonha and Mucuri (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 358.350/2013
Record Dates: First submitted 2014-03-20; First posted 2014-04-15 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Cerebral Palsy;; Dental Plaque
Keywords: Cerebral Palsy;; Toothbrushing;; Dental Plaque
MeSH Terms: conditions — Cerebral Palsy; Dental Plaque

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- manual brushing (Experimental): manual brushing; Oral-B®, Stages 4, Rio de Janeiro, Rio de Janeiro;
  Interventions: Device: manual brushing
- electric toothbrush linked (Experimental): electric toothbrush linked; Braun - Oral-B®, D2010K, Rio de Janeiro, Rio de Janeiro
  Interventions: Device: electric toothbrush linked
- off electric toothbrush (Experimental): off electric toothbrush; Braun - Oral-B®, D2010K, Rio de Janeiro, Rio de Janeiro
  Interventions: Device: off electric toothbrush

INTERVENTIONS:
Device: manual brushing — Tooth brushing
  Other Names: manual brushing; (Oral-B®, Stages 4, Rio de Janeiro, Rio de Janeiro)
  Arms: manual brushing
Device: electric toothbrush linked — Tooth brushing
  Other Names: electric toothbrush linked; Braun - Oral-B®, D2010K, Rio de Janeiro, Rio de Janeiro
  Arms: electric toothbrush linked
Device: off electric toothbrush — Tooth brushing
  Other Names: off electric toothbrush; Braun - Oral-B®, D2010K, Rio de Janeiro, Rio de Janeiro
  Arms: off electric toothbrush

SUMMARY:
The aim of the present study was to determine the effectiveness of brushing with an electric toothbrush switched on and switched off in comparison to manual brushing for the removal of dental plaque in children aged four to 16 years with cerebral palsy.

DETAILED DESCRIPTION:
Advances in the design and type of movement of electric toothbrushes can determine the increase in effectiveness in the control of biofilm by caregivers and patients.There is a paucity of studies evaluating the effectiveness of the electric toothbrush compared to manual toothbrush specifically in patients with cerebral palsy.Only one study used the electric toothbrush in patients with cerebral palsy and demonstrated superiority of the electric toothbrush over the manual. However, the study investigated the effect of various cleaning strategies on symptoms of gingival inflammation, not specifically focusing on the comparison of the efficiency of removal of biofilm from the manual toothbrush and electric toothbrush. The primary objective of this study was to evaluate the effectiveness of the electric brush on and off the removal of dental plaque in subjects with cerebral palsy compared to manual toothbrush. The secondary objective was to characterize the study as socioeconomic population.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of cerebral palsy

Exclusion Criteria:

* who did not complete the cycle three brushings

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Removal of dental plaque | after brushing three minutes duration
  Before and after brushings were assessed levels of plaque accumulation. For evaluation of the dental plaque index of Quigley-Hein plaque modified Turesky was used.
  The escovções were performed by caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Nayara Kelly Lyrio Ferraz, MsC, Principal Investigator — Federal University of the Valleys of Jequitinhonha and Mucuri
Locations (1):
- Universidade Federal dos Vales do Jequitinhonha e Mucuri, Diamantina, Minas Gerais, Brazil